CLINICAL TRIAL: NCT06004154
Title: Post-therapeutic Imaging Evaluation of Patients With Horton's Disease (Giant Cell Arteritis)
Brief Title: Post-therapeutic Imaging Evaluation of Patients With Horton's Disease (Giant Cell Arteritis) (EvHortim)
Acronym: EvHortim
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GCL_2023_3
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Injected cerebral MRI angiography and ultrasound of the superior aortic trunks, temporal and axillary arteries — Injected cerebral MRI angiography and ultrasound of the superior aortic trunks, temporal and axillary arteries added to the usual follow-up at 1, 3, 6 and 12 months

SUMMARY:
Giant cell arteritis (GCA), also known as Horton's disease, is an inflammatory arteritis of the large and medium-sized arteries, with an estimated incidence of 17.8/100,000 in people over 50.

The disease presents potential ophthalmological, neurological, cardiac and aortic vascular complications, making diagnosis an emergency in cases of suspected Horton's disease.

only corticosteroid therapy started as early as possible can prevent these complications.

Diagnosis has historically relied on temporal artery biopsy, but the recent ACR/EULAR 2022 classification criteria propose alternatives to this invasive examination, in particular imaging tests such as temporal artery ultrasound and PET scans. Although not included in these latest recommendations, high-definition wall MRI can also provide arguments in favor of this diagnosis, and avoid the need for a temporal artery biopsy, the sensitivity of which is only 75%. The investigators recently demonstrated in a prospective cohort that wall MRI, possibly coupled with temporal artery ultrasound or retinal angiography, was far superior to temporal artery biopsy in diagnostic performance.

The main limitation of these imaging tests is the lack of data in the literature on the evolution of abnormalities over time, and in particular after initiation of oral corticosteroid therapy. This uncertainty makes it difficult to use these examinations to monitor disease activity, particularly in cases of suspected relapse, a frequent situation in which the clinician is regularly put at fault due to an often frustrating symptomatology and the possible absence of a frank biological inflammatory syndrome.

The investigators propose to conduct a study aimed at describing the evolution of cranial vessel wall abnormalities on wall MRI and ultrasound by systematically repeating these examinations at 1 month, 3 months from the initial MRI performed at diagnosis, in addition to the follow-up performed as part of care at 6 and 12 months from diagnosis. In the event of a relapse in the intervening period, a new MRI scan can be performed and compared with the most recent MRI scan, to look for evidence of disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 and over
* Having received informed consent to participate in the study
* Affiliated or beneficiary of a social insurance scheme
* Patients with giant cell arteritis according to ACR/EULAR 2022 criteria
* Diagnosed with MRI and ultrasound.

Exclusion Criteria:

* Absolute or relative contraindication to MRI (incompatible implantable device, claustrophobia, etc.)
* Hypersensitivity to gadobutrol
* Patient under legal protection
* Pregnant or breast-feeding women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Fondation A de Rothschild Hospital for Horton's disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Describe the evolution over time of angiographic-MRI abnormalities at 1 month, 3 months, 6 and 12 months from the diagnosis of Horton's disease. | Day0 to Month12
  thickening (yes/no)
Describe the evolution over time of ultrasound abnormalities at 1 month, 3 months, 6 and 12 months from the diagnosis of Horton's disease. | Day0 to Month12
  contrast enhancement (yes/no)
Describe the evolution over time of ultrasound abnormalities at 1 month, 3 months, 6 and 12 months from the diagnosis of Horton's disease. | Day0 to Month12
  halo measurement (in mm)
Describe the evolution over time of ultrasound abnormalities at 1 month, 3 months, 6 and 12 months from the diagnosis of Horton's disease. | Day0 to Month12
  intima-media thickness measurement (in mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France